CLINICAL TRIAL: NCT00225680
Title: ELUTES II - In Stent ELUTES Study
Brief Title: In Stent ELUTES Study
Acronym: ELUTES II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 524
Record Dates: First submitted 2005-09-12; First posted 2005-09-26 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery; stent; drug eluting; patency; restenosis
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Device: drug eluting coronary stent

SUMMARY:
This trial will compare the long term safety and effectiveness of the V Flex Plus PTX Drug Eluting coronary stent with conventional treatment for in-stent restenosis for coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given informed consent
* Patient has target lesion in native coronary artery or coronary bypass graft
* Patient has in-stent restenosis >60%
* Patient has reference artery diameter 2.7-3.5
* Patient agrees to return for clinical assessment at 1, 6, 9, 12 and 24 months and for a treadmill test at 9 months and an angiogram at 9 months and 24 months.

Exclusion Criteria:

* Patient is less than 18 years of age
* Patient is pregnant or breast feeding
* Patient has history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Patient is simultaneously participating in another investigative interventional cardiovascular drug or device study.
* Patient has known hypersensitivity or contraindication to aspirin or stainless steel or a sensitivity to contrast agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124
Dates: Start 2002-04; Study Completion 2005-08

PRIMARY OUTCOMES:
Angiographic target vessel failure (TVF) at follow up

SECONDARY OUTCOMES:
Major adverse events
Target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ivan DeScheerder, MD, Principal Investigator — University Hospital of Gathuisberg
Locations (1):
- Contact Sponsor, Bloomington, Indiana, United States